CLINICAL TRIAL: NCT03393234
Title: Study of Safety and Feasibility of the Intersphincteric Resection With or Without Intraoperative Radiation in Low Rectal Cancer
Brief Title: Intersphincteric Resection With or Without Intraoperative Radiation in Rectal Cancer
Acronym: IDAVON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISR and IORT
Record Dates: First submitted 2018-01-01; First posted 2018-01-08 (Actual); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Rectal Cancer
Keywords: Ultra-low rectal cancer; Intersphincteric resection; IORT
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be assigned to two different groups and receive intraoperative radiation randomly. The care provider and investigator also don't know the concrete situation of the patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A group (Experimental): Patients who receive interphincteric resection (ISR) in this group will be given extra intraoperative radiation by INTRBEAM using low energy X-ray.
  Interventions: Radiation: Interoperative radiation by INTRABEAM using low energy X-ray
- B group (No Intervention): Patients who only receive interphincteric resection (ISR) in this group without intraoperative radiation.

INTERVENTIONS:
Radiation: Interoperative radiation by INTRABEAM using low energy X-ray — Intrabeam is a mobile Platform for Intraoperative Radiotherapy (IORT) produced by the ZEISS company in Germany.Interoperative radiation by INTRABEAM using low energy X-ray.The Intrabeam PRS appears to be a safe technique for delivering IORT in rectal cancer patients.
  Arms: A group

SUMMARY:
The purpose of this study was to research on the safety and feasibility of ISR combined with low energy X ray intra-operative radiotherapy for the patients with local advanced rectal cancer.

DETAILED DESCRIPTION:
Inter-sphincteric resection (ISR) has become an increasingly popular optional surgical tool for the treatment of very low rectal cancer. Nowadays, preoperative criteria for Lap ISR were the patients whose diagnosed with clinical stages T1-2 and N0_1, which only a few patients with early stages can benefit from it. However, intra-operative radiotherapy with low energy X ray applied by Intrabeam is becoming an accepted radiotherapy technique for treatment of cancers. The purpose of this study was to research on the safety and feasibility of ISR combined with low energy X ray intra-operative radiotherapy for the patients with local advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* those whom were preoperatively assessed to be in clinical stageT3 or has lymphatic metastasis by MRI or ultrasonic endoscopy;
* the lower edge of the tumor is away from the anal edge by less than 5 cm, or away from the dentate line by less than 3cm;
* in intra-operative separation, the lower edge of the tumor is below the plane of the levator ani muscle or the tumor is hard to separate;
* those in T4 stage and could be radically resected by intra-operative surgeon assessment;
* adequate preoperative sphincter function and continence; (vi)local spread restricted to the rectal wall or the IAS.
* absence of distant metastases.

Exclusion Criteria:

* clinical T4 tumors based on the Union for International Cancer Control UICC TNM classification (7th edition):
* infiltrating gross appearance of the tumors;
* poorly differentiated adenocarcinoma by biopsy specimens;
* a degree of preoperative incontinence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival | 3 years
  Compare 3-year disease free survival in patients with resectable rectal cancer treated with or without radiation.

SECONDARY OUTCOMES:
local recurrence rate | 1 years
  In our study, no matter whether distant metastases occurred, if there was the presence of any anastomotic, pelvic, or lateral node recurrences recorded by pathologic or clinical examination, we defined it as local recurrence.
R0 resection rate | 1 years
  To calculate the radical resection rate.
sphincter muscle function | 1 years
  Indicated by the anorectal manometry
anorectal manometry | 1 years
  To measure the anus pressure to indirectly reflect the sphincter muscle function
predictive biomarkers | 3 years
  Each follow-up, the biomarkers such as CEA,CA19-9 etc were recorded.
sexual function | 1 years
  Investigated by the questionnaire including the International Index of Erectile dysfunction. (IIEF5)

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
When the investigators complete the study and publish our data.
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Derived] Wang M, Xue W, Zhao Z, Li Y, Wang X, Li T, Zou Y, Song X, Zhang M, Wang T, Yang J, Wang C, Wang S. Laparoscopic intersphincteric resection with intraoperative radiotherapy using low-energy X-rays for locally advanced ultra-low rectal cancer. World J Surg Oncol. 2018 Jul 7;16(1):133. doi: 10.1186/s12957-018-1430-6. PMID 29981575